CLINICAL TRIAL: NCT04874948
Title: A Single-Center, Open Label Study to Investigate the Mass Balance, Excretion Pathways and Metabolites After a Single Oral Dose of 500 MG, 3.7 MBq, [14C]BTZ-043 in Healthy Male Volunteers
Brief Title: Absorption, Elimination and Safety of 14C-labeled Radioactive BTZ-043, a New Compound in TB Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Michael Hoelscher (Other)
Collaborators: Leibniz Institute for Natural Product Research and Infection Biology Hans Knöll Institute (Other)
Responsible Party: Sponsor-Investigator, Michael Hoelscher, Director, Ludwig-Maximilians - University of Munich
Organization: Ludwig-Maximilians - University of Munich (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LMU-IMPH-BTZ-043-03
Record Dates: First submitted 2021-04-22; First posted 2021-05-06 (Actual); Results first posted 2024-12-05 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Tuberculosis; Tuberculosis, Pulmonary; Bacterial Infections Respiratory; Lung Diseases; Mycobacterium Infections
Keywords: Anti-Bacterial Agents
MeSH Terms: conditions — Tuberculosis; Tuberculosis, Pulmonary; Lung Diseases; Mycobacterium Infections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single oral administration of 500 mg BTZ-043 containing 3.7 MBq of [14C]BTZ-043 (Experimental): 4 subjects to receive a single oral administration of 14C-labeled radioactive 500mg BTZ-043
  Interventions: Drug: 500mg BTZ-043 containing 3.7 MBq of [14C]BTZ-043

INTERVENTIONS:
Drug: 500mg BTZ-043 containing 3.7 MBq of [14C]BTZ-043 — Single oral administration of 14C-labeled radioactive 500mg BTZ-043

SUMMARY:
This study is a Phase 1, single-center, open-label study to investigate the absorption, metabolism, and excretion of BTZ-043 after a single oral administration of 500 mg BTZ-043 containing 3.7 MBq of [14C]BTZ-043 in 4 healthy adult male subjects

DETAILED DESCRIPTION:
A total of 4 evaluable subjects completing all procedures are required. Six (6) subjects will be enrolled in the cohort in order to have 4 evaluable subjects.

The study will consist of a screening period (Day -21 to -2), a baseline period (Day -1), a single dose treatment on Day 1 with a minimum of 96 hours (=4 days) post dose in-house observation period (Days -1 up to afternoon Day 5), and a follow-up visit 30 days (±2 days) after the [14C]BTZ-043 dose.

Subjects will be administered a single 500 mg [14C]BTZ-043 dose as drinking suspension. Subjects will be confined to the clinical site for at least 96 hours following drug administration (ie, afternoon of Day 5). During this time, blood, feces, and urine samples for measurement of [14C]BTZ-043 and metabolites will be collected.

The subjects will be released from the clinic approximately 96 hours to 168 hours after dose administration and upon satisfactory recovery of radioactivity (at least 90%) approved by the Sponsor's scientific advisor after consulation of the Sponsor.

ELIGIBILITY:
Inclusion Criteria:

1. Sex : male
2. Age : 18 years to 55 years, inclusive, at screening.
3. Body mass index (BMI) : 18.0 to 29.0 kg/m2, inclusive, at screening.
4. Weight : 55 to 90 kg, inclusive, at screening.
5. Status : healthy subjects.
6. Male subjects, if not surgically sterilized, must agree to use adequate contraception and not donate sperm from admission to the clinical research center until 90 days after the follow-up visit. Adequate contraception for the male subject (and his female partner, if she is of childbearing potential) is defined as using hormonal contraceptives or an intrauterine device combined with at least 1 of the following forms of contraception: a diaphragm, a cervical cap, or a condom. Total abstinence, in accordance with the lifestyle of the subject, is also acceptable.
7. All prescribed medication must have been stopped at least 30 days prior to admission to the clinical research center.
8. All over-the-counter medications, vitamin preparations (especially vitamin C), other food supplements, and herbal medications (eg, St. John's wort) must have been stopped at least 14 days prior to admission to the clinical research center. An exception is made for paracetamol, which is allowed up to 48 hours prior to study drug administration.
9. No vaccination within 14 days prior to study drug administration.
10. Ability and willingness to abstain from alcohol from 48 hours (2 days) prior to screening and admission to the clinical research center.
11. Ability and willingness to abstain from methylxanthine-containing beverages or food (coffee, tea, cola, chocolate, and energy drinks), grapefruit (juice), corn (whole corn kernels and popcorn), cruciferous vegetables, and bitter oranges from 48 hours (2 days) prior to admission to the clinical research center.
12. Good physical and mental health on the basis of medical history, physical examination, clinical laboratory, ECG, and vital signs, as judged by the Investigator.
13. Willing and able to sign the ICF.

Exclusion Criteria:

1. Participation in another study with a radiation burden of >0.1 mSv and ≤1 mSv in the period of 1 year prior to screening; a radiation burden of >1.1 mSv and ≤2 mSv in the period of 2 years prior to screening; a radiation burden of >2.1 mSv and ≤3 mSv in the period of 3 years prior to screening, etc.
2. Exposure to radiation for diagnostic reasons (except dental X-rays and plain X-rays of thorax and bony skeleton [excluding spinal column]), or during work within 1 year prior to drug administration.
3. Irregular defecation pattern (less than once per day on average).
4. Employee of PRA, Nuvisan, or the Sponsor.
5. History of relevant drug and/or food allergies.
6. Using tobacco products within 60 days prior to drug administration.
7. History of alcohol abuse or drug addiction (including soft drugs like cannabis products).
8. Positive drug and alcohol screen (opiates, methadone, cocaine, amphetamines [including ecstasy], cannabinoids, barbiturates, benzodiazepines, gamma-hydroxybutyric acid, tricyclic antidepressants, and alcohol) at screening or admission to the clinical research center.
9. Average intake of more than 24 grams of alcohol per day.
10. Positive screen for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibodies, or HIV 1 and 2 antibodies.
11. Participation in a drug study within 30 days prior to drug administration in the current study. Participation in more than 4 drug studies in the 12 months prior to drug administration in the current study.
12. Donation or loss of more than 450 mL of blood within 60 days prior to drug administration. Donation or loss of more than 1.5 liters of blood in the 10 months prior to drug administration in the current study.
13. Significant and/or acute illness within 5 days prior to drug administration that may impact safety assessments, in the opinion of the Investigator.
14. Unwillingness to consume the Food and Drug Administration (FDA)-recommended high-fat breakfast.
15. Unsuitable veins for infusion or blood sampling.
16. Positive nasopharyngeal PCR test for SARS-CoV-2 on Day -1.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2021-10-08 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Jaap van Lier, MD, Principal Investigator — PRA Health Sciences (PRA) - Early Development Services (EDS)
Locations (1):
- PRA Health Sciences (PRA) - Early Development Services (EDS), Groningen, Netherlands

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Screening started on 27th September 2021. The first participant was enrolled on October 8th, 2021. The healthy volunteers were recruited by PRA Health Sciences - Early Development Services in 9728 NZ Groningen
Groups:
- Single Oral Administration of 500 mg BTZ-043 Containing 3.7 MBq of [14C]BTZ-043: 4 subjects to receive a single oral administration of 14C-labeled radioactive 500mg BTZ-043 containing 3.7 MBq of [14C]BTZ-043
Period: Overall Study
Arm/Group | Single Oral Administration of 500 mg BTZ-043 Containing 3.7 MBq of [14C]BTZ-043
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Single Oral Administration of 500 mg BTZ-043 Containing 3.7 MBq of [14C]BTZ-043
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 22 (3)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 3
  Race: White + Black or African American | 1
Region of Enrollment [Number; unit: participants]
  Netherlands | 4
BMI [Mean (Standard Deviation); unit: kg/m²] | 24.3 (4.0)
Height [Mean (Standard Deviation); unit: cm] | 177 (2)
Weight [Mean (Standard Deviation); unit: kg] | 75.7 (13.0)

OUTCOME MEASURES:

1. Primary Outcome: Rates and Routes of Excretion
Description: To determine the rates and routes of excretion of [14C]BTZ-043-related radioactivity, including mass balance of total drug-related radioactivity in urine and feces (and vomit, if applicable), following the oral administration of a single 500 mg dose of [14C]BTZ-043 in healthy male volunteers. All excreta were collected for the analysis for 14C quick or normal counts of total radioactivity (as feasible). the radioactivity measured was translated into mg eq (Radioactivity equivalent to 1 mg BTZ-043).
Time Frame: Urine and faeces were collected from the administration of the study medication until cumulative excretion reached 90% of total radioactivity administered. This was achieved by all subjects after 168 hours.
Population: Per protocol
Measure: Mean (Standard Deviation); unit: mg eq
Arm/Group | Single Oral Administration of 500 mg BTZ-043 Containing 3.7 MBq of [14C]BTZ-043
Number analyzed (Participants) | 4
mg eq
  total drug-related radioactivity in urine | 331 (23.2)
  total drug-related radioactivity in faeces | 162 (23.0)

2. Primary Outcome: Pharmacokinetics of Total Radioactivity in Blood and Plasma (Cmax)
Description: To determine the pharmacokinetics (PK) of total radioactivity in whole blood and in plasma. Measured radioactivity was translated into ng equivalent of BTZ-043. Based on the ng eq, pharmacokinetic parameters were calculated.
Time Frame: Blood samples for total radioactivity were collected from day 1 until 168 h post dosing
Population: per protocol
Measure: Mean (Standard Deviation); unit: ng eq/mL
Arm/Group | Single Oral Administration of 500 mg BTZ-043 Containing 3.7 MBq of [14C]BTZ-043
Number analyzed (Participants) | 4
ng eq/mL
  Cmax Plasma | 8730 (2550)
  Cmax Blood | 4970 (1370)

3. Primary Outcome: Pharmacokinetics of Total Radioactivity in Blood and Plasma (AUC-t)
Description: as for outcome 2
Time Frame: Blood samples for total radioactivity were collected from day 1 until 168 h post dosing
Population: per protocol
Measure: Mean (Standard Deviation); unit: h*ng eq/mL
Arm/Group | Single Oral Administration of 500 mg BTZ-043 Containing 3.7 MBq of [14C]BTZ-043
Number analyzed (Participants) | 4
h*ng eq/mL
  AUC-t Plasma | 125000 (26900)
  AUC-t Blood | 76700 (18500)

4. Primary Outcome: Pharmacokinetics of Total Radioactivity in Blood (T1/2)
Description: as for outcome 2
Time Frame: Blood samples for total radioactivity were collected from day 1 until 168 h post dosing
Population: per protocol. On participant excluded as value was justed unreliable
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Single Oral Administration of 500 mg BTZ-043 Containing 3.7 MBq of [14C]BTZ-043
Number analyzed (Participants) | 3
h | 158 (24.7)

5. Primary Outcome: Pharmacokinetics of Total Radioactivity in Plasma (T1/2)
Description: as for outcome 2
Time Frame: Blood samples for total radioactivity were collected from day 1 until 168 h post dosing
Population: per protocol.
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Single Oral Administration of 500 mg BTZ-043 Containing 3.7 MBq of [14C]BTZ-043
Number analyzed (Participants) | 4
h | 186 (18.9)

6. Primary Outcome: Plasma PK of BTZ-043 and Main Metabolites (Cmax)
Description: To characterize the plasma PK of BTZ-043 and main metabolites by liquid chromatography-mass spectrometry (LC-MS), if applicable. BTZ-043 is metabolized in the human body. Some of the metabolites were known prior to this study like the main metabolite M2, a hydrid Meisenheimer complex or the aminometabolite M1. Metabolite M4 and M10 were known before as well, therefore, the bioanalytical methods mentioned above could be developed and validated for these metabolites.Pharmacokinetic parameters are calculated from the individual plasma level measurements.
Time Frame: Day 1 to Day 3
Population: Per protocol
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Single Oral Administration of 500 mg BTZ-043 Containing 3.7 MBq of [14C]BTZ-043
Number analyzed (Participants) | 4
ng/mL
  Cmax BTZ-043 | 1600 (509)
  Cmax M1 | 163 (27.5)
  Cmax M2 | 5180 (1310)
  Cmax M4total | 1190 (455)
  Cmax M10 | 30.6 (6.50)

7. Primary Outcome: Plasma PK of BTZ-043 and Main Metabolites (AUC-last)
Description: To characterize the plasma PK of BTZ-043 and main metabolites by liquid chromatography-mass spectrometry (LC-MS), if applicable. BTZ-043 is metabolized in the human body. Some of the metabolites were known prior to this study like the main metabolite M2, a hydrid Meisenheimer complex or the aminometabolite M1. Metabolite M4 and M10 were known before as well, therefore, the bioanalytical methods mentioned above could be developed and validated for these metabolites. Pharmacokinetic parameters are calculated from the individual plasma level measurements.
Time Frame: Day 1 to Day 3
Population: Per protocol
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Single Oral Administration of 500 mg BTZ-043 Containing 3.7 MBq of [14C]BTZ-043
Number analyzed (Participants) | 4
h*ng/mL
  AUClast BTZ-043 | 3920 (842)
  AUClast M1 | 2710 (433)
  AUClast M2 | 41000 (6220)
  AUClast M4total | 10300 (3990)
  AUClast M10 | 505 (199)

8. Primary Outcome: Plasma PK of BTZ-043 and Main Metabolites (t1/2)
Description: as for outcome 7
Time Frame: Day 1 to Day 3
Population: Per protocol
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Single Oral Administration of 500 mg BTZ-043 Containing 3.7 MBq of [14C]BTZ-043
Number analyzed (Participants) | 4
h
  T1/2 BTZ-043 | 2.43 (1.01)
  T1/2 M1: number analyzed (Participants) | 1
  T1/2 M1 | 8.65 (0)
  T1/2 M2 | 4.90 (0.591)
  T1/2 M4total | 3.83 (0.281)
  T1/2 M10 | 18.9 (10.2)

9. Primary Outcome: Urine Concentrations of BTZ-043 and Main Metabolites
Description: Urine volume was measured after every micturation and hamilton pools have been prepared for analysis of BTZ-043 and main metabolites by LC-MS. BTZ-043 could only be measured in urine within the first 24h, then no additional BTZ-043 was excreted in urine anymore. The same applies for M1. M2, M4 total and M10 total excretion could be measured in urine up to 48h post dose.
Time Frame: Assessed from time of dosing up to 168 h post dose. BTZ-043 and metabolites were excreted fom 0 - 24 h (BTZ-043 and M1) and from 0 - 48 h (M2, M4 total and M10 total).
Population: Per protocol
Measure: Mean (Standard Deviation); unit: mg eq
Arm/Group | Single Oral Administration of 500 mg BTZ-043 Containing 3.7 MBq of [14C]BTZ-043
Number analyzed (Participants) | 4
mg eq
  BTZ-043 (M0) Cumulative Amount Excreted 0 - 24h | 8.83 (4.51)
  M1 Cumulative Amount Excreted 0 - 24h | 1.53 (0.518)
  M2 Cumulative Amount Excreted 0 - 24h | 53.9 (17.1)
  M2 Cumulative Amount Excreted 0 - 48h | 54.7 (17.3)
  M4 total Cumulative Amount Excreted 0 - 24h | 59.4 (9.77)
  M4 total Cumulative Amount Excreted 0 - 48h | 60.5 (10.2)
  M10 total Cumulative Amount Excreted 0 - 24h | 2.47 (1.33)
  M10 total Cumulative Amount Excreted 0 - 48h | 2.65 (1.45)
  Sum(M0, M1, M2, M4total, M10) Cumulative Amount Excreted 0-24h | 126 (15.7)
  Sum(M0, M1, M2, M4total, M10) Cumulative Amount Excreted 0-48h | 128 (16.4)

10. Secondary Outcome: Number of Adverse Events
Description: To assess the safety and tolerability of a single 500 mg oral dose of BTZ-043 administered to healthy volunteers.
Time Frame: Day -1 to day 32
Population: Received at least one dose of BTZ-043
Measure: Number; unit: Adverse Events
Arm/Group | Single Oral Administration of 500 mg BTZ-043 Containing 3.7 MBq of [14C]BTZ-043
Number analyzed (Participants) | 4
Adverse Events | 6

ADVERSE EVENTS:
Time Frame: Day -1 (admission) until follow-up on day 31 or 32
Description: An AE is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medical treatment or procedure that may or may not be considered related to the medical treatment or procedure. AE definitions according to ICH topic E2A.
  All AEs reported or apparent from their physical appearance during the clinical study were reported on the AE eCRF page.
  Severity of AEs was graded using the most current version of the MedDRA
Arm/Group | Single Oral Administration of 500 mg BTZ-043 Containing 3.7 MBq of [14C]BTZ-043
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 4/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Oral Administration of 500 mg BTZ-043 Containing 3.7 MBq of [14C]BTZ-043 (N=4)
Dizziness (Nervous system disorders) | 4 (4)
Somnolence (Nervous system disorders) | 1 (1)
Oral Herpes (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-07-01): https://cdn.clinicaltrials.gov/large-docs/48/NCT04874948/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-02): https://cdn.clinicaltrials.gov/large-docs/48/NCT04874948/SAP_001.pdf